CLINICAL TRIAL: NCT07046663
Title: Long-term Assessment of Chlormethine Gel in Mycosis Fungoides: A Multicenter Retrospective Cohort Study
Brief Title: Long-term Assessment of Chlormethine Gel in Mycosis Fungoides
Acronym: FIL_CLOR-CTCL
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Other Study IDs: FIL_CLOR-CTCL
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Cutaneous T-Cell Lymphoma/Mycosis Fungoides
Keywords: mycosis fungoides; cutaneous T-cell lymphoma; chlormethine gel; long term assessment
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who started treatment with chlormethine gel, from September 1, 2019 to September 30, 2024

SUMMARY:
The study aims to provide comprehensive insights into the long-term therapeutic outcomes, potential adverse effects, and overall patient experience with chlormethine gel, thereby informing clinical practice and guiding future treatment strategies for mycosis fungoides.

DETAILED DESCRIPTION:
Primary cutaneous lymphomas (PCLs) are a rare group of lymphoproliferative disorders with neoplastic lymphocyte proliferation in the skin. Cutaneous T-cell lymphomas (CTCL) make up 75% of PCLs, with mycosis fungoides (MF) being the most common. The cause of MF is unclear, but persistent antigenic stimulation and chronic inflammation may lead to neoplastic transformation. Pathogenesis involves genetic and epigenetic abnormalities, with a crucial role played by the skin microenvironment. Data from the International PROCLIPI registry (PROspective Cutaneous Lymphoma International Prognostic Index Validation and Evaluation) provide insight into the clinical management and outcomes of CTCL. This study has confirmed that early-stage disease has a relatively favorable prognosis, with a 5-year survival rate of about 90% for stage IA patients. Treatment is stage-dependent. Early stages are managed with skin-directed therapies (topical steroids, chlormethine and phototherapy) as first lines, while refractory or advanced disease requires systemic therapies such as interferon, bexarotene, and extracorporeal photopheresis. Chemotherapy and new monoclonal agents are used for refractory advanced cases. Topical chlormethine (TC) is an alkylating agent successfully used in treating CTCL since the 1950s. It works by a cytotoxic mechanism on DNA, altering the growth of neoplastic cells and enhancing the host's immunogenic potential. Initially, TC was packaged in an aqueous solution, but its use was limited by a high rate of skin hypersensitivity. In 2013, a multicenter, randomized, blinded phase II study compared 0.02% TC ointment with 0.02% TC gel, demonstrating the gel's non-inferiority to the ointment. The study also recorded longer and faster responses in the gel arm. No detectable systemic absorption of the drug was observed in patients' blood, consistent with previous case series. The evidence on the development of secondary neoplasms is controversial, particularly the risk of non-melanoma skin cancers (NMSC), which ranges from 0 to 9%. This risk is higher in patients previously treated with other modalities known to increase skin cancer incidence (e.g., radiotherapy and phototherapy). Melanoma development was reported by Ramsay et al. in a single patient with Fitzpatrick type I skin and a history of NMSC.

Real-world data from numerous studies have confirmed the efficacy of TC gel in treating early-stage MF and its use in combination with systemic therapies for advanced stages. In particular, the PROVE study, based on US real-world experience, demonstrated that modulating the TC schedule to every other day maintained good efficacy while reducing the incidence of adverse events, such as irritant contact dermatitis (ICD), and improving patient compliance. In a previous retrospective study on the first patients treated with TC gel in Italy, was showed that hyperpigmentation correlates with good response.

Currently, there is a lack of data on long-term response, recurrence rates after initial response, and the effect on treated areas considering the significant irritative response.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 18
* Histologically confirmed diagnosis of MF based on WHO Classification of Tumours, Haematolymphoid Tumours, 5th edition
* Patients who are capable of understanding and willing, and able to read and write in Italian
* Patients who have signed informed consent form
* Patients who started treatment with chlormethine gel, from September 1, 2019 to September 30, 2024.
* Patients must have a minimum follow-up period of 6 months following the initiation of chlormethine treatment.
* Availability of complete medical records in order to provide protocol required variables.

Exclusion Criteria:

* Patients for whom retrospective data or information on the type of therapy, duration, and clinical outcomes are not available in the center's medical records.
* Refuse to sign a written informed consent.
* Patients not meeting the above-mentioned inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with histologically confirmed MF treated with TC gel (from September 1, 2019 to September 30, 2024) at the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of complete remission (rate CR) | Up to 12 months
  Rate of complete remission (rate CR) according to CAILS and mCAILS tools and mSWAT after 6 months from the start of treatment

SECONDARY OUTCOMES:
Percentage of CR and ORR (CR+PR) | Up to 12 months
  Percentage after 3, 6 and 12 months from start of treatment of CR and ORR (CR+PR)
Nelson-Aalen estimation | Up to 12 months
  Nelson-Aalen estimation from start of treatment to first attained CR
Kaplan-Meier estimation of Time to recurrence (TTR) | Up to 12 months
  Kaplan-Meier estimation of Time to recurrence (TTR) from date of attained CR
Percentage of relevant toxicities over an extended use | Up to 12 months
  Percentage of relevant toxicities over an extended use
Percentages of toxicity in specific areas | Up to 12 months
  Percentages of toxicity in specific areas (face and skin folds)
Percentages of skin toxicity by patient characteristics | Up to 12 months
  Percentages of skin toxicity by patient characteristics
Frequency of use of different regimens | Up to 12 months
  Frequency of use of different therapy regimens

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Alberti Violetti, Principal Investigator — UOC Dermatologia - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milano, Italy
Locations (20):
- Italy (20):
  - AOU Ospedali Riuniti - Clinica di Ematologia, Ancona
  - SC Dermatologia, ASST-Papa Giovanni XXIII,, Bergamo
  - UO Dermatologia - IRCCS Policlinico S.Orsola-Malpighi, Bologna
  - UO Dermatologia ASST Spedali Civili Brescia, Brescia
  - UOC di Dermatologia - Azienda Ospedaliero-Universitaria di Cagliari, presidio Ospedaliero S. Giovanni di Dio, Cagliari
  - UOC Dermatologia - Azienda Ospedaliero Universitaria Policlinico "G. Rodolico - San Marco", Catania
  - UOC Ematologia - ARNAS Nuovo Ospedale Garibaldi Nesima, Catania
  - S.C. Dermatologia, AUSL Toscana Centro e Università degli Studi di Firenze, Presidio Ospedaliero Palagi, Florence
  - SC Dermatologia, Ente Ospedaliero Ospedali Galliera di Genova, Genova
  - UO Dermatologia, ASST-Lecco, Azienda Ospedaliera A. Manzoni, Lecco
  - UO Dermatologia Clinica - IRCCS Ospedale San Raffaele di Milano, Milan
  - UOC Dermatologia - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - UOC Clinica Dermatologica - AOU "Luigi Vanvitelli", Napoli
  - SCDU Dermatologia; AOU Maggiore della Carità di Novara, Novara
  - SC Dermatologia - Fondazione IRCCS Policlinico San Matteo Clinica Dermatologica, Pavia
  - UOSD Porfirie e Malattie rare - Istituto Dermatologico San Gallicano- IRCCS, Roma
  - UO Dermatologia - IRCCS Humanitas, Rozzano
  - SC Dermatologia U - AOU Città della Salute e della Scienza di Torino, Torino
  - UOC Dermatologia e Venerologia - ASP Trapani, PO Sant'Antonio Abate, Trapani
  - UOC Dermatologia - Azienda Ospedaliera Universitaria Integrata di Verona, Verona